CLINICAL TRIAL: NCT06943651
Title: Empowering Healthy Lifestyle Behaviour Through Personalized Intervention Portfolios to Prevent and Control Obesity in Young Adults - A Pilot Study
Brief Title: Empowering Healthy Lifestyle Behavior to Prevent and Control Obesity in Young Adults
Acronym: HW8YAPilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Elsa Lamy, Principal Investigator, Head of the Laboratory of Oral Biology and Salivary Proteomics of MED, University of Evora, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UEVHealthyW8YAdults; GA - 101080645 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2024-11-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Obese; Overweight
Keywords: Obesity; Overweight; Digital twin; Obesity prevention; Lifestyle
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: This is a longitudinal study, non-controlled. Participants will receive the developed healthy life-style recommender solution for the duration of the study, and endpoints within subjects will be compared before and after.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test of healthyW8 Digital Twin of healthy lifestyle recommendations (Experimental): Individuals will have access to a digital tool, putting together nutrition, physical activity and emotional aspects. Participant interaction with the tool, through registration collected or inputed by the individual will allow personalized recommendations.
  Interventions: Device: HealthyW8 Digital Twin of healthy lifestyle recommendations

INTERVENTIONS:
Device: HealthyW8 Digital Twin of healthy lifestyle recommendations — The applied intervention with the developed healthy lifestyle recommender system will be unique and is not used in any other clinical study. However, a large number of intervention studies on young adults' obesity, considering nudging (e.g. 60 in www.clinical.trials.gov), were found. Among the registered clinical trials in the referred database, 3 considered young adults obesity and saliva salivary analysis, but with a different purpose. Moreover, the type of digital solution that will be tested will put together different aspects that are not usually to see together in the same application. These different lifestyle aspects will be used for personalized recommendations.

SUMMARY:
This human study will be a pilot trial that will precede a planned more long-term intervention trial. It will focus on young adults (age 18 to 25 y). The main purpose is to study whether the healthy lifestyle recommender solution, reflecting a multi-portfolio intervention and developed within this project, is well accepted by the participants, has a decent adherence (i.e. user time of the app), and whether the overall design is well suited to the participants, in order that they will improve dietary habits. This study will be of longitudinal design without a control group.

At present, numbers of persons with overweight and obesity continue to grow in most countries worldwide. Young adults are at risk since in in this period of life most people start to be independent from their families, with the consequent decisions about their food and lifestyle choices. It is frequent that at this time an increase in irregularity of meals and unhealthy food choices, occurs, together with changes in physical activity habits and social or individual pressures. Because of this, it is essential to give tools to these individuals that will allow them to make healthy choices and to have healthy habits, since they will be the future adult population that will raise and inspire the next generation. As solutions to combat the trend toward increasing overweight and obesity are much in need, the present study aims to intervene with the developed healthy lifestyle recommender solution to address various factors known to constitute a risk for developing obesity, including socio-demographic aspects, psychological/behavioural ones, physical activity, dietary patterns, among other. Such a multi-dimensional portfolio approach is believed to be very much needed for the prevention of obesity and co-morbidities, and the personalization of the solution, as well as the nudging/gamification.

DETAILED DESCRIPTION:
The applied intervention with the developed healthy lifestyle recommender system will be unique and is not used in any other clinical study. However, a large number of intervention studies on young adults' obesity, considering nudging (e.g. 60 in www.clinical.trials.gov), were found. Among the registered clinical trials in the referred database, 3 considered young adults obesity and saliva salivary analysis.

The investigators judge the risk for the participant as low, since only saliva will be collected which collection is totally non-invasive. The administered intervention is expected to be effective, based on the multi-level nature of the tools applied.

This is a longitudinal study, non-controlled. Participants will receive the developed healthy life-style recommender solution for the duration of the study, and endpoints within subjects will be compared before and after.

The investigators are aware of the potential influence of seasons and other longitudinal changes on the outcomes, however as the endpoints are rather motivation and adherence, the investigators deem the design as appropriate. Moreover, in case of salivary parameters, which can be more sensitive to this type of variation, the collection in three successive days, before and at the end of the trial (to be analysed as pooled samples) will minimize these potential effects.

The intervention is the developed eHealth solution, i.e. the healthy lifestyle recommender system. It is based on a previously developed meal recommender system, but will be much extended, resulting in a multilevel portfolio intervention regarding:

1. Suggesting personalized meal recommendations,
2. Proposing physical activities tailored to the individuals' capabilities and preferences,
3. Measuring and considering emotional and psychological parameters,
4. Proposing additional healthy life-style patterns regarding e.g. sleeping patterns, alcohol and tobacco consumption, engaging in social activities etc.

The detailed nature of the interventions will first be developed during co-creation and then targeted to the participating individual. The intervention will include collecting urinary and saliva samples, as well as measuring anthropometrics and collecting data (personal, socio-demographics, general health and well-being, physical activity and eating patterns, among other) via questionnaires.

The study duration will be 3 months from the official start to the end. Following a first interview to test participants eligibility, the investigators have compiled a list of exemplary endpoints in the following, providing an overview about the sampling frequency.

Young adults (age 18-25 y) will be recruited via university and local hospital (Hospital do Espirito Santo - Évora), with help from the researchers from the School of Health Sciences, by direct advertisement and by recommendation of Hospital dietitians. The run-in time of the study will be long enough to assure recruitment of the required number of persons. The participants will be followed up regularly by phone-calls from the team of the University of Évora (e.g. weekly), and via contact maintained through the developed healthy lifestyle recommender solution. Should recruitment be insufficient, additional advertisement via local newspapers will be carried out, and the run-in time be extended.

Participants will receive the developed healthy lifestyle recommender solution. The individuals will then make use of the healthy lifestyle recommender solution for the entire study, i.e. a personalized, multi-level portfolio intervention will be tailored to the individual. The details of this intervention, including also nudges and gamification aspects will have to be developed during the project (WPs 2). Weekly phone-calls with participants from both groups will assure further adherence to the study.

Collected samples (month 0 and month 3) will be stored locally at University of Evora. All data and questionnaires will be collected by trained personnel, using RedCap platform. Data will be stored under a protected server, under the responsibility of Luxemburg Institute of Health, which is the leading institution of the project HealthyW8, under which this study is being developed. Individual data will be not linked to participants identification, since each participant will receive a code, at the beginning, answering all questionnaires and collecting all the samples under that identification (code). Only the researcher responsible for the study will have assess to the correspondence between identification and codes. This correspondence will be stored in an external drive, safely stored in the University of Evora and without being connected to internet.

The intervention will only require the healthy lifestyle recommender solution in form of an app. In addition, participants in the intervention arm will be able to access the Open Stakeholders Platform to access further information on healthy living. All data collected will be compiled in clinical report forms that will be generated by the University of Evora team. Saliva will be collected by trained researchers from the University of Evora. Regarding questionnaires, the investigators will use previous developed and validated questionnaires, such as the IPAQ questionnaire for physical activity or the SF-36 questionnaire for healthy lifestyle.

ELIGIBILITY:
Inclusion criteria:

* To be young adult (age 18-25 y)
* To reside in Portugal
* To be overweight (BMI between 25-30 kg/m2)
* Women and men

Exclusion Criteria:

* To have a manifest chronic diseases (e.g. cancer)
* To be already in energy restriction or following a specific diet (on their own or advised by their physician)
* To have eating behavior pathologies.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to digital tool | 3-month
  Adherence time to the lifestyle recommender solution, in order to determine the success of application of the healthy-lifestyle recommender solution to the target population (the young adults).
Satisfaction relative to the digital solution | 3 months
  The satisfaction for the use of the digital solution will be assessed through questionnaires addressing the user-friendliness and limitation or problems encountered.
  Scales will be used, where higher scores mean higher satisfaction.

SECONDARY OUTCOMES:
Anthropometry | 3-month
  Secondary outcomes (measured at the end of the 3-month period of the pilot):
  Change of BMI, relatively to the beginning of the intervention.
Fat Mass | 3-months
  Reduction of fat mass will be determined by measuring body composition through bio impedance at beginning and end of 3-month trial. The difference will allow to assess if fat mass decreased or increased, during this period.
Blood Pressure | 3-month
  Blood pressure (systolic, diastolic) will be measured at the beginning and at the end of the 3-month trial.
Salivary biomarkers | 3-month
  Saliva composition will be assessed for measuring concentration of C-reactive protein, salivary IgA, glucose and insulin. This will be done at the beginning and at the end of the 3-month trial, to assess changes during this period.
Salivary markers of stress | 3-month
  Concentrations of salivary cortisol will be measured at the beginning and at the end of the 3-month period of the trial.
Salivary Amylase | 3-month
  The enzymatic activity per unit of saliva volume will be assessed for amylase. This will be done in saliva collected at the beginning and at the end of 3-month trial.
Physical activity | At the beginning of the study
  The level of physical-activity habits will be assessed using the IPAQ short form. The participants will be assessed at the beginning of the trial.
Diet | 1 week
  The dietary habits will be assessed using a 24h-recall, applied for 3 different days, at the beginning of the trial. The results will allow to estimate the average amount of macro- and micronutrients daily ingested.

OTHER OUTCOMES:
Antropometric data | 3-month
  Height and body weight will be measured to calculate BMI, both at beginning and at the end of 3-month period.

IPD SHARING:
Plan to Share IPD: Yes
The investigators will follow the General Data Protection Regulation (EU) 2016/679 of 27 April 2016 (known as the GDPR) and all subsequent texts replacing or supplementing this Regulation Before the start of the study, all subjects will be informed about the aim of the study, the study protocol, as well as risks/benefits.
  Only the researcher responsible for the study will have access to the correspondence between identification and the codes generated. This correspondence will be stored in a computer protected with password, not linked to internet and in a drive, stored in the University of Evora. All data (questionnaires, samples, etc.) will be identified with the participant code and not personal identification. Data will be presented treated, and no individual data, that could allow participant identification, will be public presented.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the beginning until the final of HealthyW8 project (from 2025-2028)
Access Criteria: Only the researcher responsible for the study will have access to the correspondence between identification and codification. All the other researchers will have access only to codified individual data. Individual data will be shared only with the researchers responsible for statistical analysis and not public presented.